CLINICAL TRIAL: NCT04822792
Title: Pan-cancer Early-stage Detection by Liquid Biopsy in Peripheral Blood: a Multi-center, Prospective Observational Study
Brief Title: Pan-canceR Early-Stage deteCtion by lIquid Biopsy tEchNique projecT
Acronym: PRESCIENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RSCD2020002
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Cancer
Keywords: Cancer; Liquid biopsy; Cell-free DNA (cfDNA); Early detection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer Arm: Participants with new diagnosis of cancer, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test
- Benign Diseases Arm: Participants with benign diseases corresponding to the tumor types in the Cancer Arm, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test
- Healthy Arm: Participants without known presence of malignancies or benign disease, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test

INTERVENTIONS:
Device: Multi-cancer early detection test — Blood collection and multi-cancer early detection test

SUMMARY:
PRESCIENT is a multi-center, prospective observational study aimed to detect cancers early by combined assays for serum protein markers and cell-free DNA (cfDNA) methylation markers. Blood RNA markers will also be evaluated. The study will enroll approximately 11879 participants, including participants with malignancies or benign diseases, and healthy participants.

ELIGIBILITY:
Inclusion Criteria for All the Participants:

* Ability to provide a written informed consent
* 40-75 years old

Exclusion Criteria for All the Participants:

* Inability to comply with study procedures
* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer

Inclusion Criteria for Cancer Arm Participants:

* Confirmed diagnosis or suspicious cases of one of the 22 types of malignancies within 42 days prior to study blood draw
* No prior or ongoing anti-cancer therapy (local or systematic) prior to study blood draw

Exclusion Criteria for Cancer Arm Participants:

* Known prior diagnosis of malignancies
* Other current malignant diseases or multiple primary tumors
* No confirmed diagnosis of cancer by histopathological or radiological assessments within 42 days of study blood draw, or diagnosis of a benign disease by histopathological assessments, or inability to characterize whether the lesion is malignant or benign
* Non-small-cell lung cancer patients with ground-class nodularity by radiological examination

Inclusion Criteria for Benign Diseases Arm Participants:

* Confirmed diagnosis of benign diseases corresponding to the tumor types in the Cancer Arm by histopathological or radiological assessments within 90 days prior to study blood draw
* No prior treatment of benign diseases prior to study blood draw

Exclusion Criteria for Benign Diseases Arm Participants:

* History of malignancies
* Current malignancies or precancerous lesions
* No confirmed diagnosis of a benign disease by radiological, endoscopic or histopathological assessments within 42 days of study blood draw, or inability to characterize whether the lesion is malignant or benign

Inclusion Criteria for Non-tumor (Healthy) Arm Participants:

* No cancer-related symptoms or discomfort within 30 days prior to study blood draw
* No clinically significant finding by LDCT or ultrasound
* No clinically significant finding by breast ultrasound or Molybdenum Target Mammography Detection, or Thinprep cytologic test (TCT) detection for female participants
* No active hepatitis B or hepatitis C infection

Exclusion Criteria for Non-tumor (Healthy) Arm Participants:

* Prior or ongoing treatment of cancer within 3 years prior to study blood draw
* Clinically significant or uncontrolled comorbidities

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be re recruited from medical centers and assigned into three arms, including participants with new diagnosis of malignancies or corresponding benign diseases, and participants without the presence of malignancies or benign diseases.
Sampling Method: Non-Probability Sample
Enrollment: 11879 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of early detection of 22 types of cancers and Tissue of origin (TOO) accuracy of a cfDNA methylation-based model, in combination with serum tumor markers | 22 months

SECONDARY OUTCOMES:
Sensitivity and specificity of a cfDNA methylation-based model combined with serum tumor markers in participants with cancers or benign diseases | 22 months
Sensitivity and specificity of serum tumor markers, cfDNA methylation-based model, and a cfDNA methylation-based model combined with serum tumor markers, in participants with cancers and healthy participants | 22 months
Sensitivity and specificity of early detection of cancer in different stages | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, M.D., Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No